CLINICAL TRIAL: NCT03928353
Title: A Phase 2A, Randomized, Double-blind, Placebo-controlled, Single Dose, Sequential Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PB2452 With Ticagrelor Pretreatment in Older and Elderly Subjects and With High-Dose Ticagrelor Pretreatment in Healthy Younger Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, PK and PD of PB2452 in Healthy Younger, Older and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SFJ Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB2452-PT-CL-0002
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Aftercare

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1: 18 g PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for a total of 5 doses
  Interventions: Drug: Ticagrelor Oral Tablet - Pre-Treatment; Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride
- 2: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg+90 mg BID for a total of 5 doses
  Interventions: Drug: Ticagrelor Oral Tablet - Pre-Treatment; Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride
- 3: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment
- 4: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride With Ticagrelor Oral Tablet: 180 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment
- 5: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx) (Experimental): PB2452 Infusion or Placebo - Sodium Chloride with Ticagrelor Oral Tablet: 180 mg BID for a total of 5 doses
  Interventions: Drug: PB2452 Infusion; Drug: Placebo - Sodium Chloride; Drug: Ticagrelor Oral Tablet - Pre-Treatment; Drug: Ticagrelor Oral Tablet - Pre-Treatment and Post-Treatment

INTERVENTIONS:
Drug: PB2452 Infusion — 30 minute - 24 hour infusion
  Arms: 3: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 4: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 5: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: Placebo - Sodium Chloride — 30 minute - 24 hour infusion
  Arms: 3: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 4: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 5: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: Ticagrelor Oral Tablet - Pre-Treatment — Ticagrelor 180 mg + 90 mg BID for 5 doses prior to PB2452 or Placebo
  Arms: 1: 18 g PB2452 or Placebo (Ticagrelor Pre-Trx); 2: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 5: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: Ticagrelor Oral Tablet - Pre-Treatment and Post-Treatment — Ticagrelor 180 mg + 90 mg BID for 5 doses prior to PB2452 or Placebo and Ticagrelor 180 mg 24 hours following PB2452 or Placebo
  Arms: 5: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: Ticagrelor Oral Tablet - Pre-Treatment — Ticagrelor 180 mg BID for 5 doses prior to PB2452 or Placebo
  Arms: 3: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 4: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx); 5: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: PB2452 Infusion — 30 minute - 16 hour infusion
  Arms: 1: 18 g PB2452 or Placebo (Ticagrelor Pre-Trx); 2: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)
Drug: Placebo - Sodium Chloride — Placebo - Sodium Chloride
  Arms: 1: 18 g PB2452 or Placebo (Ticagrelor Pre-Trx); 2: 18 g or greater PB2452 or Placebo (Ticagrelor Pre-Trx)

SUMMARY:
This is a Phase 2A, randomized, double-blind, placebo-controlled, single dose, sequential group study to evaluate the safety, tolerability, PK, and PD of PB2452 vs matching placebo with ticagrelor (with or without acetylsalicylic acid (ASA)) pretreatment when various dose levels and administration regimens are administered to healthy younger (ages 18 to 50), older (ages 50 to 64 years) and elderly (ages 65 to 80 years) male and female subjects.

Up to 5 dose levels and/or administration regimens will be evaluated in up to 5 cohorts. Each cohort will include approximately 8 to 12 subjects randomized in a 3:1 ratio (PB2452:placebo).

DETAILED DESCRIPTION:
The study will consist of a Screening period, a Check-in day and Pretreatment Period, an on-site Randomization/Treatment day, 3 days on-site for treatment and safety monitoring, a Follow-up Visit (Day 7), and a Final Follow-up visit (Day 28). Seven days prior to Randomization, subjects in Cohorts 1 and 2 will be administered acetylsalicylic acid (ASA) 81 mg orally once daily (QD) until the final dose on the morning of Day 1 before receiving study drug. A ticagrelor 180 mg oral dose will be administered on the morning of Day -2 followed by either 90 mg or 180 mg every 12 hours (BID) until the 5th dose has been administered on the morning of Day 1.

On Day 1, subjects who meet all the inclusion criteria and none of the exclusion criteria will be randomized in a ratio 3:1 (PB2452:placebo), to receive an IV dose of PB2452 or placebo 2 hours following the 5th ticagrelor dose. Subjects may be discharged from the clinical site between Days 3 and 7 inclusive and will return for a Follow-up visit on Day 7, if already discharged, and on Day 28 (±2 days).

ELIGIBILITY:
Inclusion Criteria:

1. The subject provides written informed consent and agrees to comply with all protocol requirements.
2. The subject is male or female between 18 and 80 years of age, inclusive (50 to 80 years for Cohorts 1-2, 18 to 50 years for Cohorts 3-5).
3. The subject has a body mass index (BMI) between 18 and 35 kg/m2 and a weight of ≥50 kg but ≤120 kg, inclusive, at Screening.
4. The subject is considered by the investigator to be in good general health, as determined by medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination findings at Screening. Older and elderly subjects with chronic, stable, and well-controlled medical conditions are eligible provided they meet all other inclusion/exclusion criteria. Some examples of stable and well-controlled medical conditions include but are not limited to:

   * Hypertension (HTN) controlled with ≤2 antihypertensive drugs
   * Diabetes controlled with diet/exercise or treated with up to 2 oral diabetes medications
   * Subjects with diabetes must have a glycated hemoglobin HbA1c ≤8 mg/dL at Screening.
   * Mild hepatic enzyme elevation (aspartate aminotransferase (AST) or alanine transaminase (ALT) <1.5 x ULN or total bilirubin <1.2 x ULN)
   * Controlled hyperlipidemia (defined with a Screening low density lipoprotein LDL <160 mg/dL)
5. Specific inclusionary laboratory values at Screening and Check-in require:

   * White blood cell (WBC) count, platelet count, hemoglobin (Hgb) level within normal range, as defined by the clinical laboratory
   * Thyroid stimulating hormone (TSH) level within normal range, as defined by the clinical laboratory at Screening
   * Prothrombin time (PT) and partial thromboplastin time (PTT) level within normal range, as defined by the clinical laboratory
6. Subjects taking medications for well-controlled medical conditions must have been on a stable dose (meaning no changes in dose) for at least 30 days prior to Screening visit.
7. Older and elderly subjects entering the study who are not already taking daily ASA must be willing to start an 81 mg daily dose of ASA on Day -7 and continue daily dosing until the final dose is administered on the morning of Day 1. Subjects entering the study who are already taking ASA daily will be administered 81 mg ASA daily between Day -7 and Day 1 and must suspend further ASA dosing until discharge from the clinical facility.
8. Female subjects of childbearing potential must not be pregnant, lactating, or planning to become pregnant for 3 months after the last dose of study drug, and have a negative serum pregnancy test at Screening and Check-in. Female subjects of childbearing potential must use 2 effective methods of birth control from 30 days before study drug administration through to the end of the study.

   * Effective birth control methods include oral, implantable, patch, or injectable contraceptive hormone treatment, hormone-containing intrauterine device that has been in place ≥2 months prior to Screening, sponge, diaphragm, or cervical cap with spermicidal gel or cream for female subjects or condom or vasectomy for male subjects.
   * Women are considered to not be of childbearing potential if they have fulfilled one of these criteria: documentation of irreversible surgical sterilization (i.e., hysterectomy or bilateral oophorectomy [not tubal ligation]) or are postmenopausal (defined as amenorrhea for 12 consecutive months following cessation of all exogenous hormonal treatments, and documented plasma follicle-stimulating hormone (FSH) level >40 IU/mL) or amenorrhea for 24 consecutive months.
   * Male subjects with partners of childbearing potential must agree to use appropriate and effective measures of contraception (e.g., condom plus diaphragm with spermicide, condom plus spermicide) during the study and for 30 days after the last dose of study drug, and refrain from donating sperm for ≥90 days following the last dose of study drug.

Exclusion Criteria:

1. Concern the subject may be unable to comply with study procedures and/or follow up, or, in the opinion of the investigator, the subject is not suitable for entry into the study
2. History of any acute or chronic medical disorder expected to decrease the life expectancy of the subject
3. History or presence of gastrointestinal (GI), hepatic (with the exception of Gilbert's syndrome), or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
4. Significant renal insufficiency, as indicated by estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 according to the Modification of Diet in Renal Disease (MDRD) equation
5. Any clinically significant (CS) acute illness, medical/surgical procedure, or trauma within 4 weeks of administration of study drug or any planned surgical procedure that will occur during the study (from Screening through the Day 28 [±2 days] Follow-up visit)
6. Any CS abnormal findings in physical examination, vital signs, laboratory assessments, and ECG parameters identified during Screening or Check-in. Note: abnormal results may be repeated for confirmation immediately after the first out of range measurement. Abnormal vital signs may be repeated twice if needed, immediately after the first abnormal result and/or after the subject has rested for at least 10 minutes.

   Specific vital sign exclusionary criteria occurring after 10 minutes of supine rest are any of the following:
   * Systolic blood pressure (SBP) <100 or >160 mm Hg
   * Diastolic blood pressure (DBP) <40 or >95 mm Hg
   * Resting heart rate (HR) <50 or >100 beats per minute (bpm)

   Specific exclusionary criteria for ECG parameters at Screening or Check-in include any of the following:
   * Prolonged Fridericia-corrected QT interval (QTcF) >450 milliseconds (msec)
   * Shortened QTcF <340 msec, or pause >3 seconds
   * Family history of long QT syndrome
7. Any specific contraindication to Brilinta® as described in the Brilinta® prescribing information and:

   * History of intracranial hemorrhage, active bleeding, or hypersensitivity or allergic reaction to ticagrelor or any component of the product
   * Any history of severe head trauma, intracranial neoplasm, arteriovenous malformation, aneurysm, or proliferative retinopathy
   * Any history of intraocular, retroperitoneal, or spinal bleeding
   * Have taken, within 30 days of Screening, any oral or parenteral anticoagulant, including low molecular-weight heparin
   * Stool sample testing positive for occult blood within 3 months of Screening or at any time during the Screening Period
8. Receiving chronic treatment with nonsteroidal anti-inflammatory drugs (NSAIDS; [including ASA >100 mg daily]), anticoagulants, or other antiplatelet agents that cannot be discontinued 14 days prior to randomization (including clopidogrel, prasugrel, ticlopidine, dipyridamole, or cilostazol)
9. Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at Screening
10. Concomitant oral or IV therapy with strong cytochrome P450 3A4 (CYP3A) inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers, which cannot be stopped within at least 5 half-lives, but not fewer than 10 days, before randomization
11. Consumption of grapefruit or grapefruit juice, Seville orange or Seville orange containing products (e.g., marmalade), or xanthine containing products within 48 hours before dosing with study drug
12. Prescription or over the counter (OTC) medications within 14 days before the first dose of study drug unless specifically allowed by protocol. (Permitted medications include multivitamins, paracetamol [up to 2g per day], and/or treatments for chronic stable diseases, provided the drug and dose have been stable for ≥30 days prior to administration of study drug)
13. Has received another investigational drug (defined as a small molecule or biologic compound which has not been approved for marketing) within 30 days of the administration of study drug in this study or within 5 half-lives of the prior study drug, whichever is longer
14. Positive test result for alcohol or drugs of abuse at Screening or Check-in
15. Participated in strenuous activity or contact sports within 24 hours before the infusion of study drug or while confined in the clinical site
16. History of severe or ongoing allergy/hypersensitivity to any drug or biologic therapeutic agent
17. Involvement with any previous Sponsor's or study site employee or their close relatives (e.g., spouse, parents, siblings, or children whether biological or legally adopted)
18. Previously received PB2452 or had been randomized to receive study drug in an earlier cohort for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LuAnn Bundrant, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, younger, older, and elderly male and female participants were enrolled and randomized in a single center.
Groups:
- Part A - Cohort 1: Older and elderly participants pretreated with ticagrelor + ASA received 18 g of PB2452 intravenously (IV) during the treatment period.
- Part A - Cohort 2: Older and elderly participants pretreated with ticagrelor + ASA received 18 g of PB2452 IV during the treatment period. Following completion of Cohort 1, the previous Sponsor instructed the clinical site to administer study drug in the same manner as in Cohort 1 in Cohort 2.
- Part A - Placebo (Pooled): Older and elderly participants pretreated with ticagrelor + ASA received 0.9% sodium chloride IV during the treatment period.
- Part B - Cohort 3: Healthy and younger participants pretreated with a high dose of ticagrelor (180 mg BID) received 36 g of PB252 IV during the treatment period.
- Part B - Placebo: Healthy and younger participants pretreated with a high dose of ticagrelor (180 mg BID) received 0.9% sodium chloride IV during the treatment period.
Period: Overall Study
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Started | 6 | 5 | 4 | 6 | 2
Completed | 6 | 5 | 4 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and randomized in the study.
Groups:
- Part A - Cohort 1; Part A - Cohort 2: Older and elderly participants pretreated with ticagrelor + ASA received 18 g of PB2452 IV during the treatment period.
- Part A - Placebo: Older and elderly participants pretreated with ticagrelor + ASA received 0.9% sodium chloride IV during the treatment period.
- Total: Total of all reporting groups
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Placebo | Part B - Cohort 3 | Part B - Placebo | Total
Number analyzed (Participants) | 6 | 5 | 4 | 6 | 2 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (7.24) | 63.8 (9.31) | 60.5 (4.65) | 34.7 (8.14) | 30.5 (2.12) | 51.48 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 1 | 1 | 11
  Male | 2 | 2 | 2 | 5 | 1 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population of participants based on their ethnicity.
  Participants
    Hispanic or Latino | 3 | 0 | 1 | 1 | 1 | 6
    Not Hispanic or Latino | 3 | 5 | 3 | 5 | 1 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population of participants based on their race.
  Participants
    Black or African American | 2 | 2 | 0 | 3 | 0 | 7
    White | 4 | 3 | 4 | 3 | 2 | 16
Renal Function [Count of Participants; unit: Participants]
  Mild (Mild decrease in kidney function) | 3 | 5 | 2 | 2 | 1 | 13
  Normal (Normal kidney function) | 3 | 0 | 2 | 4 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Treatment-emergent Adverse Events (TEAEs) And Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug-related. A TEAE is defined as any AE not present before exposure to study drug or any AE already present that worsens in intensity or frequency after exposure to study drug. An SAE/suspected unexpected serious adverse reaction if, in the view of either the investigator or Sponsor, it results in any of the following outcomes: death, life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or congenital anomaly or birth defect. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Day -3 up to Day 28
Population: All participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - Cohort 1-2 (Pooled): Older and elderly participants pretreated with ticagrelor + ASA received 18 g of PB2452 IV during the treatment period.
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Participants
  TEAEs | 1 | 2 | 3 | 3 | 4 | 1
  SAEs | 0 | 1 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Number of participants with clinically significant abnormal laboratory findings for hematology, coagulation, serum chemistry, and urinalysis.
Time Frame: Day -45 up to Day 28
Population: All participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 4 | 6 | 2
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Mean Diastolic Blood Pressure at Baseline
Time Frame: Baseline
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
mmHg | 74.17 (8.42) | 67.60 (7.44) | 71.18 (8.33) | 75.25 (3.40) | 63.83 (5.91) | 61.50 (2.12)

4. Primary Outcome: Percent Change In Diastolic Blood Pressure From Baseline To Day 28
Description: Diastolic blood pressure measurements were measured at specific time points.
Time Frame: Day 1 (10, 20, 30, 45, and 60 minutes post-dose), Day 2, Day 3, Day 7, and Day 28
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Percent change in DBP
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Percent change in DBP
  Change from Baseline - Day 1/ 10 Minutes Postdose: number analyzed (Participants) | 4 | 4 | 8 | 2 | 6 | 2
  Change from Baseline - Day 1/ 10 Minutes Postdose | -2.50 (9.15) | -1.75 (5.91) | -2.13 (7.14) | -4.00 (9.90) | 4.00 (6.69) | 2.50 (7.78)
  Change from Baseline - Day 1/ 20 Minutes Postdose: number analyzed (Participants) | 6 | 4 | 10 | 3 | 6 | 2
  Change from Baseline - Day 1/ 20 Minutes Postdose | -4.33 (5.65) | -4.75 (0.96) | -4.50 (4.25) | -5.67 (1.53) | 3.50 (8.83) | 1.00 (8.49)
  Change from Baseline - Day 1/ 30 Minutes Postdose: number analyzed (Participants) | 6 | 5 | 11 | 2 | 6 | 2
  Change from Baseline - Day 1/ 30 Minutes Postdose | -3.17 (8.33) | -3.80 (2.59) | -3.45 (6.12) | -2.00 (2.83) | 9.00 (3.35) | 5.50 (3.54)
  Change from Baseline - Day 1/ 45 Minutes Postdose | -2.00 (2.53) | -3.20 (4.76) | -2.55 (3.56) | -2.00 (7.39) | 3.83 (7.68) | 0 (9.90)
  Change from Baseline Day 1/ 1 Hour Postdose | -3.67 (9.16) | 0.40 (6.58) | -1.82 (7.99) | -4.25 (9.98) | 4.67 (4.68) | 3.50 (13.44)
  Change from Baseline - Day 2/ 24 Hour | -6.17 (8.54) | -7.40 (4.62) | -6.73 (6.74) | -8.50 (6.03) | -3.33 (4.68) | 1.50 (3.54)
  Change from Baseline - Day 3/ 48 Hour | -5.67 (14.39) | -3.20 (5.63) | -4.55 (10.86) | -7.75 (10.81) | 2.67 (6.89) | -1.00 (8.49)
  Change from Baseline - Day 7 | -6.00 (9.88) | 0.40 (6.91) | -3.09 (8.89) | -9.00 (6.68) | 6.50 (5.58) | 7.50 (7.78)
  Change from Baseline - Day 28 | 4.67 (9.54) | 0.40 (5.94) | 2.73 (8.04) | -3.75 (12.31) | 5.17 (7.31) | 10.00 (4.24)

5. Primary Outcome: Mean Systolic Blood Pressure at Baseline
Time Frame: Baseline
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
mmHg | 128.33 (17.15) | 115.40 (11.08) | 122.45 (15.55) | 119.00 (17.80) | 113.14 (8.75) | 108.50 (0.71)

6. Primary Outcome: Percent Change In Systolic Blood Pressure From Baseline To Day 28
Description: Systolic blood pressure measurements were measured at specific time points.
Time Frame: Day 1 (10, 20, 30, 45, and 60 minutes post-dose), Day 2, Day 3, Day 7, and Day 28
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Percent change in SBP
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Percent change in SBP
  Change from Baseline - Day 1/ 10 Minutes Postdose: number analyzed (Participants) | 4 | 4 | 8 | 2 | 6 | 2
  Change from Baseline - Day 1/ 10 Minutes Postdose | -6.75 (4.11) | 0.75 (5.85) | -3.00 (6.16) | -7.50 (20.51) | 5.83 (7.31) | 2.00 (11.31)
  Change from Baseline - Day 1/ 20 Minutes Postdose: number analyzed (Participants) | 6 | 4 | 10 | 3 | 6 | 2
  Change from Baseline - Day 1/ 20 Minutes Postdose | -7.67 (13.98) | 2.75 (9.18) | -3.50 (12.87) | -6.33 (4.93) | 2.83 (5.81) | -0.50 (0.71)
  Change from Baseline - Day 1/ 30 Minutes Postdose: number analyzed (Participants) | 6 | 5 | 11 | 2 | 6 | 2
  Change from Baseline - Day 1/ 30 Minutes Postdose | -5.33 (14.07) | -0.20 (4.09) | -3.00 (10.62) | -5.50 (9.19) | -0.33 (4.63) | 2.50 (9.19)
  Change from Baseline - Day 1/ 45 Minutes Postdose | -7.33 (12.88) | -3.80 (4.15) | -5.73 (9.65) | -2.25 (12.12) | 4.00 (5.59) | 3.50 (9.19)
  Change from Baseline Day 1/ 1 Hour Postdose | -8.00 (11.47) | 5.20 (14.31) | -2.00 (13.97) | 1.00 (20.05) | 0.67 (5.89) | -0.50 (12.02)
  Change from Baseline - Day 2/ 24 Hour | -14.00 (16.14) | -5.60 (10.24) | -10.18 (13.83) | -2.75 (13.52) | -2.33 (5.99) | 6.00 (1.41)
  Change from Baseline - Day 3/ 48 Hour | -17.17 (14.41) | -4.00 (10.89) | -11.18 (14.09) | -9.00 (10.36) | 2.00 (4.10) | 1.50 (3.54)
  Change from Baseline - Day 7 | -6.33 (13.87) | 2.80 (14.55) | -2.18 (14.27) | -12.00 (12.73) | 6.67 (12.48) | 3.00 (7.07)
  Change from Baseline - Day 28 | 1.50 (15.14) | 9.80 (10.96) | 5.27 (13.47) | 0 (10.92) | 9.67 (5.68) | 12.50 (4.95)

7. Primary Outcome: Mean Oral Body Temperature at Baseline
Time Frame: Baseline
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Degrees Celcius | 36.17 (0.34) | 35.88 (0.15) | 36.04 (0.30) | 36.25 (0.24) | 36.20 (0.38) | 36.35 (0.07)

8. Primary Outcome: Percent Change In Oral Body Temperature From Baseline To Day 28
Description: Body temperature measurements were measured at specific time points.
Time Frame: Day 1 (45 and 60 minutes post-dose), Day 2, Day 3, Day 7, and Day 28
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Percent change in oral body temperature
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Percent change in oral body temperature
  Change from Baseline - Day 1/ 45 Minutes Postdose: number analyzed (Participants) | 6 | 4 | 10 | 4 | 6 | 2
  Change from Baseline - Day 1/ 45 Minutes Postdose | 0.18 (0.53) | 0 (0.14) | 0.11 (0.41) | 0.15 (0.34) | 0.13 (0.23) | -0.10 (0.28)
  Change from Baseline Day 1/ 1 Hour Postdose | -0.10 (0.32) | 0 (0.21) | -0.05 (0.27) | 0.15 (0.26) | 0.20 (0.17) | 0.10 (0.42)
  Change from Baseline - Day 2/ 24 Hour | 0.05 (0.35) | 0.10 (0.29) | 0.07 (0.31) | 0.10 (0.32) | -0.03 (0.43) | -0.05 (0.07)
  Change from Baseline - Day 3/ 48 Hour | -0.05 (0.50) | 0.24 (0.05) | 0.08 (0.39) | 0.25 (0.17) | 0.17 (0.14) | 0 (0.28)
  Change from Baseline - Day 7 | 0.02 (0.34) | 0.44 (0.29) | 0.21 (0.38) | 0.07 (0.19) | 0.25 (0.29) | 0 (0.28)
  Change from Baseline - Day 28 | -0.33 (0.34) | 0.34 (0.15) | -0.03 (0.44) | -0.15 (0.19) | 0.30 (0.23) | -0.35 (0.35)

9. Primary Outcome: Mean Respiratory Rate at Baseline
Time Frame: Baseline
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Breaths per minute | 14.33 (1.51) | 13.60 (2.61) | 14.00 (2.00) | 12.50 (2.52) | 15.67 (2.94) | 17.00 (1.41)

10. Primary Outcome: Percent Change In Respiratory Rate From Baseline To Day 28
Description: Respiratory rate measurements were measured at specific time points.
Time Frame: Day 1 (45 and 60 minutes post-dose), Day 2, Day 3, Day 7, and Day 28
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Percent change in respiratory rate
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Percent change in respiratory rate
  Change from Baseline - Day 1/ 45 Minutes Postdose: number analyzed (Participants) | 6 | 4 | 11 | 4 | 6 | 2
  Change from Baseline - Day 1/ 45 Minutes Postdose | -3.33 (1.63) | 0.50 (3.79) | -1.80 (3.19) | -0.50 (3.00) | -1.00 (2.10) | -3.00 (1.41)
  Change from Baseline Day 1/ 1 Hour Postdose | -2.00 (1.26) | -0.40 (3.85) | -1.27 (2.72) | 1.00 (2.58) | -4.33 (3.44) | -4.00 (2.83)
  Change from Baseline - Day 2/ 24 Hour | -0.67 (3.27) | 2.40 (2.19) | 0.73 (3.13) | 1.50 (1.91) | -1.00 (3.29) | -4.00 (2.83)
  Change from Baseline - Day 3/ 48 Hour | -2.00 (2.19) | 0.40 (3.29) | -0.91 (2.88) | 0.50 (1.00) | -2.67 (2.07) | -3.00 (1.41)
  Change from Baseline - Day 7 | -0.33 (2.66) | 0.40 (2.61) | 0 (2.53) | 1.00 (1.15) | -2.00 (2.53) | -1.00 (1.41)
  Change from Baseline - Day 28 | -0.33 (3.44) | 0.80 (3.35) | 0.18 (3.28) | 1.00 (2.00) | -3.67 (4.08) | -6.00 (2.83)

11. Primary Outcome: Mean Heart Rate at Baseline
Time Frame: Baseline
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Beats per minute | 70.17 (8.04) | 60.20 (5.89) | 65.64 (8.56) | 63.00 (10.74) | 65.50 (5.21) | 78.00 (29.70)

12. Primary Outcome: Percent Change In Heart Rate From Baseline To Day 28
Description: Heart rate measurements were measured at specific time points.
Time Frame: Baseline, Day 1 (10, 20, 30, 45, and 60 minutes post-dose), Day 2, Day 3, Day 7, and Day 28
Population: All participants who received any amount of study drug.
Measure: Mean (Standard Deviation); unit: Percent change in heart rate
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Percent change in heart rate
  Change from Baseline - Day 1/ 10 Minutes Postdose: number analyzed (Participants) | 4 | 4 | 8 | 2 | 6 | 2
  Change from Baseline - Day 1/ 10 Minutes Postdose | -5.25 (11.24) | 0.50 (6.61) | -2.38 (9.07) | -4.00 (7.07) | -3.17 (6.68) | -16.00 (21.21)
  Change from Baseline - Day 1/ 20 Minutes Postdose: number analyzed (Participants) | 6 | 4 | 10 | 3 | 6 | 2
  Change from Baseline - Day 1/ 20 Minutes Postdose | -4.17 (9.41) | -0.50 (3.79) | -2.70 (7.59) | 0 (9.85) | -3.17 (3.19) | -11.50 (16.26)
  Change from Baseline - Day 1/ 30 Minutes Postdose: number analyzed (Participants) | 6 | 5 | 11 | 2 | 6 | 2
  Change from Baseline - Day 1/ 30 Minutes Postdose | -4.50 (8.53) | -1.20 (4.60) | -3.00 (6.91) | -0.50 (9.19) | -4.83 (5.95) | -7.50 (24.75)
  Change from Baseline - Day 1/ 45 Minutes Postdose | -3.83 (8.54) | -1.80 (4.44) | -2.91 (6.74) | 2.25 (4.50) | -3.83 (4.36) | -9.00 (18.38)
  Change from Baseline Day 1/ 1 Hour Postdose | -3.17 (8.50) | 0 (5.15) | -1.73 (7.03) | 1.75 (7.41) | -2.67 (4.72) | -13.00 (18.38)
  Change from Baseline - Day 2/ 24 Hour | -1.17 (10.46) | 1.40 (3.78) | 0 (7.89) | 5.25 (3.20) | -0.33 (6.50) | -12.50 (17.68)
  Change from Baseline - Day 3/ 48 Hour | -3.50 (8.64) | 1.80 (6.69) | -1.09 (7.93) | 2.25 (5.74) | -1.00 (4.94) | -12.50 (12.02)
  Change from Baseline - Day 7 | -1.67 (9.07) | 5.40 (5.68) | 1.55 (8.23) | 0 (12.19) | -4.00 (5.55) | -15.50 (21.92)
  Change from Baseline - Day 28 | -5.17 (7.52) | 1.40 (6.62) | -2.18 (7.59) | -1.75 (13.62) | -4.33 (6.59) | -18.00 (24.04)

13. Primary Outcome: Incidence Of Clinically Significant 12-Lead Electrocardiogram (ECG) Findings
Description: Number of participants per cohort with clinically significant ECG findings.
Time Frame: Up to Day 28
Population: All participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 4 | 6 | 2
Participants | 0 | 1 | 0 | 0 | 0

14. Primary Outcome: Participants Experiencing Anti-drug Antibodies (ADAs)
Description: Number of participants who developed ADAs to PB2452.
Time Frame: Day -3, Day 1, Day 7, and Day 28
Population: All participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Cohort 1-2 (Pooled) | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 11 | 4 | 6 | 2
Participants
  Day -3 | 2 | 0 | 2 | 0 | 0 | 0
  Day 1 | 0 | 0 | 0 | 0 | 0 | 0
  Day 7 | 2 | 0 | 2 | 0 | 1 | 0
  Day 28 | 2 | 0 | 2 | 0 | 1 | 0

15. Primary Outcome: Number of Participants With Adverse Events During Physical Examination
Description: Participants with adverse events noted during physical exam between baseline and end of study.
Time Frame: Baseline through Day 28
Population: All participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - Cohort 2: Older and elderly participants pretreated with ticagrelor + ASA received 18 g of PB2452 IV during the treatment period. Following completion of Cohort 1, the Sponsor instructed the clinical site to administer study drug in the same manner as in Cohort 1 in Cohort 2.
Arm/Group | Part A - Cohort 1 | Part A - Cohort 2 | Part A - Placebo (Pooled) | Part B - Cohort 3 | Part B - Placebo
Number analyzed (Participants) | 6 | 5 | 4 | 6 | 2
Participants | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day -3 (Pretreatment) up to Day 28
Groups:
- Part A - Cohort 1: 18 g PB2452 (ASA + Ticagrelor Pre-Trx); Part A - Cohort 2: 18 g PB2452 (ASA + Ticagrelor Pre-Trx): ASA + Ticagrelor Oral Tablet - Pre-Treatment: ASA 81 mg and Ticagrelor 180 mg + 90 mg BID for 5 doses prior to PB2452 administration
  PB2452 Infusion: initial administration of 6 g bolus infused over 10 minutes followed by 6 g infused over the next 4 hours, followed by 6 g infused over the next 12 hours for a total of a 16-hour and 10 minutes infusion.
- Part A - Cohorts 1-2 Placebo: (ASA + Ticagrelor Pre-Trx): Placebo - 0.9% Sodium Chloride
  ASA + Ticagrelor Oral Tablet - Pre-Treatment: ASA 81 mg and Ticagrelor 180 mg + 90 mg BID for 5 doses prior to PB2452 administration
  Placebo - Sodium Chloride: initial administration of 6 g bolus infused over 10 minutes followed by 6 g infused over the next 4 hours, followed by 6 g infused over the next 12 hours for a total of a 16-hour and 10 minutes infusion.
- Part B - Cohort 3: 36 g PB2452 (Ticagrelor Pre-Trx): Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg BID for 5 doses prior to PB2452 administration
  PB2452 Infusion: initial administration of 12 g bolus infused over 10 minutes followed by 12 g infused over the next 6 hours, followed by 12 g infused over 18 hours for a total of 24-hour and 10 minutes infusion.
- Part B - Cohort 3 Placebo: (Ticagrelor Pre-Trx): Placebo - 0.9% Sodium Chloride
  Ticagrelor Oral Tablet - Pre-Treatment: Ticagrelor 180 mg BID for 5 doses prior to PB2452 administration
  Placebo - Sodium Chloride: initial administration of 12 g bolus infused over 10 minutes followed by 12 g infused over the next 6 hours, followed by 12 g infused over 18 hours for a total of 24-hour and 10 minutes infusion.
Arm/Group | Part A - Cohort 1: 18 g PB2452 (ASA + Ticagrelor Pre-Trx) | Part A - Cohort 2: 18 g PB2452 (ASA + Ticagrelor Pre-Trx) | Part A - Cohorts 1-2 Placebo: (ASA + Ticagrelor Pre-Trx) | Part B - Cohort 3: 36 g PB2452 (Ticagrelor Pre-Trx) | Part B - Cohort 3 Placebo: (Ticagrelor Pre-Trx)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/4 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5 | 0/4 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 1/6 | 2/5 | 3/4 | 4/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Cohort 1: 18 g PB2452 (ASA + Ticagrelor Pre-Trx) (N=6) | Part A - Cohort 2: 18 g PB2452 (ASA + Ticagrelor Pre-Trx) (N=5) | Part A - Cohorts 1-2 Placebo: (ASA + Ticagrelor Pre-Trx) (N=4) | Part B - Cohort 3: 36 g PB2452 (Ticagrelor Pre-Trx) (N=6) | Part B - Cohort 3 Placebo: (Ticagrelor Pre-Trx) (N=2)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Cohort 1: 18 g PB2452 (ASA + Ticagrelor Pre-Trx) (N=6) | Part A - Cohort 2: 18 g PB2452 (ASA + Ticagrelor Pre-Trx) (N=5) | Part A - Cohorts 1-2 Placebo: (ASA + Ticagrelor Pre-Trx) (N=4) | Part B - Cohort 3: 36 g PB2452 (Ticagrelor Pre-Trx) (N=6) | Part B - Cohort 3 Placebo: (Ticagrelor Pre-Trx) (N=2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT03928353/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03928353/SAP_001.pdf